CLINICAL TRIAL: NCT03571113
Title: Cardiac Arrest Survival Score (CRASS) - a Tool to Predict Good Neurological Outcome After Out of Hospital Cardiac Arrest
Brief Title: Cardiac Arrest Survival Score (CRASS)
Acronym: CRASS
Status: Completed | Type: Observational
Sponsor: German Resuscitation Registry (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1
Record Dates: First submitted 2018-06-16; First posted 2018-06-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest, OHCA survival score, predicting survival, German Resuscitation Registry
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development: The study population was divided into two parts by random: development dataset (5,775) and validation dataset (1,457)
  Interventions: Other: Survival / not survival
- Validation: The study population was divided into two parts by random: development dataset (5,775) and validation dataset (1,457)
  Interventions: Other: Survival / not survival

INTERVENTIONS:
Other: Survival / not survival — Outcome with good neurological status vs. bad neurological status at hospital discharge

SUMMARY:
Survival following cardiopulmonary resuscitation (CPR) from out-of-hospital cardiac arrest (OHCA) depends on numerous prehospital and in-hospital variables and interventions. The aim of this study was to develop a score to predict the resuscitation outcome after OHCA at hospital discharge.

All patients suffered OHCA between 01.01.2010 and 31.12.2016 with ROSC or ongoing CPR at hospital admission in Emergency Medical Service (EMS) systems with good quality in documentation in the German Resuscitation Registry (GRR) were included. The study population was divided into development dataset (5,775) and validation dataset (1,457) by random. Binary logistic regression analysis was used to derive the score. Hospital discharge with good neurological function (CPC 1-2 or mRS 0-2) was used as dependent variable, and various combination of potential predictor variables were used to create the model.

DETAILED DESCRIPTION:
This study is a retrospective analysis of 8,603 prospectively documented OHCA patients between 01.01.2010 and 31.12.2016 within the German Resuscitation Registry (GRR),4 attended by EMS. The GRR represents currently approximately 160 emergency medical systems who record data on out-of-hospital resuscitation attempts throughout Germany, thus encompassing approximately 30 million citizens (total population of Germany counts 85 million).

The German Resuscitation Registry for out-of-hospital cardiac arrest is divided into two different datasets:

1. The 'Preclinical care' dataset originated from the Utstein-style template aiming at documentation of pre-hospital logistic issues, presumed aetiology, resuscitation therapy and patient's initial outcome including 118 variables.12
2. The 'Postresuscitation care' dataset is aimed at documentation of in-hospital post-resuscitation efforts. The participating hospitals can choose between a basic version which includes the use of coronary angiography, temperature management and the status at hospital discharged and an extended version. This includes 156 variables and inquires especially the status at admission, initial blood gas analysis, temperature management, coronary angiography and survival at 24h after cardiac arrest, 30 days and at hospital discharge exactly.12 Participation in the registry is voluntary. The participating emergency medical services and hospitals submit their data anonymously into a central database via a web-based application. Multiple plausibility checks have been implemented into this application in order to improve data quality. The registry is organised and funded by the German Society of Anaesthesiology and Intensive Care Medicine (DGAI).

ELIGIBILITY:
Inclusion Criteria:

* OHCA between 01.01.2010 and 31.12.2016
* ROSC or ongoing CPR on hopsital admission
* high quality documentation with more than 75% documentation of post resuscitation care in hospital
* Patients cases documented in German Resuscitation Registry

Between 01.01.2010 and 31.12.2016 the 'Preclinical care' dataset contained 8,603 out-of-hospital CA patients with return of spontaneous circulation (ROSC) or ongoing CPR at hospital admission in EMS systems with good documentation quality. Good quality of documentation was defined by documented post-resuscitation care in more than 75%.

Exclusion Criteria:

* incomplete dataset
* age less than 18 years
* unknown initial ECG
* unknown age
* unknown neurological status on hospital discharge

1,371 patients were excluded from further analysis because of incomplete data in terms of age, neurological status at hospital discharge, unknown initial EKG or age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between 01.01.2010 and 31.12.2016 the 'Preclinical care' dataset contained 8,603 out-of-hospital CA patients with return of spontaneous circulation (ROSC) or ongoing CPR at hospital admission in EMS systems with good documentation quality.
Sampling Method: Non-Probability Sample
Enrollment: 8603 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
good neurological outcome | 30 days after OHCA
  CPC 1 and 2 or mRS 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Thorsten Gräsner, MD, Study Director — Institute for Emergency Medicine, Department of Anesthesiology and Intensive Care Medicine, University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grasner JT, Meybohm P, Lefering R, Wnent J, Bahr J, Messelken M, Jantzen T, Franz R, Scholz J, Schleppers A, Bottiger BW, Bein B, Fischer M; German Resuscitation Registry Study Group. ROSC after cardiac arrest--the RACA score to predict outcome after out-of-hospital cardiac arrest. Eur Heart J. 2011 Jul;32(13):1649-56. doi: 10.1093/eurheartj/ehr107. Epub 2011 Apr 22. PMID 21515626